CLINICAL TRIAL: NCT01797575
Title: A Double-blind Randomized Placebo-controlled Study of Aspirin and N-acetyl Cysteine as Adjunctive Treatments for Bipolar Disorder Patients (SMRI 11T-009)
Brief Title: N-Acetyl Cysteine and Aspirin as an Adjunctive Treatment for Bipolar Disorder
Acronym: SMRI-Bipolar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jair Soares, Professor & Chairman - PSY-Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-12-0046; SMRI (Other Grant/Funding Number: The Stanley Medical Research Institute); SMRI#11T-009 (Other Grant/Funding Number: The Stanley Medical Research Institute)
Record Dates: First submitted 2012-06-08; First posted 2013-02-22 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Mood Disorder; Bipolar Depression; Mood Swings
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Aspirin; Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Aspirin (Active Comparator): research subject will be taking aspirin 1000mg (2 capsules of 500mg) every morning in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations
  Interventions: Drug: Aspirin
- N-acetyl-cysteine (Active Comparator): research subject will be taking N-acetyl-cysteine (NAC) 1000mg (2 capsules of 500mg) two times a day in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations
  Interventions: Dietary Supplement: N-acetyl-cysteine (NAC)
- Aspirin and NAC (Active Comparator): research subject will be taking aspirin 1000mg (2 capsules of 500mg) every morning and NAC 1000mg (2 capsules of 500mg) two times a day in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations.
  Interventions: Drug: Aspirin; Dietary Supplement: N-acetyl-cysteine (NAC)
- Sugar Pill (Placebo Comparator): research subject will be taking 4 capsules of matching sugar pill( placebo) in the morning and 2 capsules of matching placebo in the evenings in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Aspirin — aspirin 1000mg (2 capsules of 500mg) every morning in addition to his/her antidepressant and/or mood stabilizer medicine
  Other Names: Ecotrin; Bayer Aspirin; Bufferin; Acetylsalicylic Acid
  Arms: Aspirin; Aspirin and NAC
Dietary Supplement: N-acetyl-cysteine (NAC) — taking N-acetyl-cysteine (NAC) 1000mg (2 capsules of 500mg) two times a day in addition to his/her antidepressant and/or mood stabilizer medicine
  Other Names: Acetylcysteine; N-Acetyl Cysteine; NAC
  Arms: Aspirin and NAC; N-acetyl-cysteine
Drug: Sugar Pill — research subject will be taking placebo in addition to his/her antidepressant and/or mood stabilizer medicine
  Arms: Sugar Pill

SUMMARY:
We propose to conduct a double-blind placebo-controlled trial with a widely available and prototypical non-steroidal anti-inflammatory agent, aspirin, and an antioxidant agent, NAC, involving symptomatic Bipolar Disorder type I and II patients having a depressive or mixed episode currently. This will be the first controlled study to test the hypothesis that aspirin and NAC, by themselves or in combination, will be beneficial in treating depression in bipolar disorder patients and in promoting mood stabilization.

Our study has the following Aims:

Aim I - Examine efficacy of aspirin in treating depression in bipolar patients in a double-blind placebo-controlled add-on design; Aim II - Examine efficacy of NAC in treating depression in bipolar patients in a double-blind placebo-controlled add-on design; Aim III - Examine efficacy of combined treatment with aspirin and NAC looking for synergistic, potentiating effects; Aim IV - Examine the role of markers of neuroinflammation, as possible mediators or modulators in therapeutic response in the treatment of depression in patients with Bipolar Disorder.

DETAILED DESCRIPTION:
study design: BD type I or II patients (n=160), on a depressive or mixed episode, who were on therapeutic doses of any of the commonly utilized mood stabilizing agents (lithium, anticonvulsants, atypical antipsychotics) for at least one month and who were still symptomatic (MADRAS >20) will be enrolled. Patients will be randomly assigned to orally receive one of 4 conditions: aspirin 1000 mg (2 capsules of 500 mg) qam, NAC 1000 mg (2 capsules of 500 mg) bid, combined aspirin and NAC at same doses as given individually or matched placebo, as an add-on medication to their ongoing treatment regimen, for an 16-week double-blind trial. After the first 8 week of the double blind treatment, the responders will keep taking the same study drug, whichever it is. And the non-responders will be re-randomized for one of the other three groups of study drugs they haven't tried yet.

Procedures to be used:

The study will be carried out at the outpatient clinics affiliated with the UT Health Science Center at Houston. After signing informed consent, patients will be submitted initially to a structure psychiatric diagnostic interview(SCID-I) to confirm the psychiatric diagnosis, followed by a physical examination and routine labs (CBC, liver function tests, electrolytes, kidney functions tests, thyroid function tests, urinalyses) to rule out relevant medical problems. Physically healthy BD patients on psychotropic medications or combinations will be enrolled and randomly assigned to receive, orally, aspirin 1000 mg qam, NAC 1000 mg bid, combination of aspirin 1000 mg qam and NAC 1000 mg bid, or placebo. The study drugs doses will remain the same for the duration of the study.

If patients qualify for the study initially based on SCID-I interview, physical examination, and routine labs (CBC, liver functions tests, electrolytes, kidney function tests, thyroid function tests, and urinalyses), but are not currently taking an approved psychotropic medication or combinations they are eligible to participate in a lead-in phase. This phase would be starting at their screening visit and last approximately 6 to 8 weeks depending on the patient's mood. During this lead-in phase, either the PI or Co-PI will evaluate the patient and prescribe either Lithium or Depakote. The patient will be monitored during this treatment phase by the PI or Co-PI and will return after two weeks for an evaluation. The evaluation will include the Columbia-Suicide Severity Rating Scale(CSSR-S) to assess risk of suicide, the Montgomery-Asberg Depression Rating Scale(MADRAS) to assess the severity of depression and the UKU side effects rating scale. If the patient is prescribed lithium, their lithium levels will be tested. The patient will continue to follow up every two weeks. At the 4 week visit, the patient will also come in for evaluation (CSSR-S MADRAS and UKU side effects rating scale).

At the 6 week visit, the patient will be re-evaluated for the double-blind study trial. If the patient has been on an adequate dose of the psychotropic medication for at least 4 weeks and score greater than 20 on the Montgomery-Asberg Depression Rating Scale (MADRS), then they will be enrolled.

If they do not meet inclusion criteria at the week 6 lead-in phase visit, they will return at Week 8 and be re-evaluated. PI and Co-PI will continue to prescribe the psychotropic medication throughout the lead-in phase (up to 8 weeks) and through the trial (up to 16 weeks).

During the lead-in phase participants will not be compensated. They will receive a voucher for their parking for each visit. They will be responsible for filling and paying for all prescriptions in both the lead-in phase and through the trial (up to 16 weeks).

Upon completion of the first 8-week double-blind trial, patients who responded to the active medication will continued on the same study drug for an additional 8 week double-blind treatment. The non-responders to one of the study drugs will be re-randomized for one of the other three groups of study not received and will remain in treatment for an additional 8 week double-blind treatment. Treatment response will be defined as improvement in the MADRS scores of at least 50%.

During the first 8-week trial, patients will be seen at weeks 0, 1, 2, 3, 4, 6 and 8 for clinical assessment and mood ratings. During the continuation trial, they will be seen at weeks 8, 10, 12, 14 and 16.

Routine labs (CBC, liver function tests, electrolytes, kidney functions tests, thyroid function tests, urinalyses) will be repeated at week 8 and week 16.

The main outcome measure for the study will be the scores on the Montgomery-Asberg Depression Rating Scale, MADRAS, which assess the severity of depressive symptoms. All patients will also be assessed with the Young Mania Rating Scale, YMRS,which assess the severity of manic symptoms. the Clinical Global Impression-Bipolar version,severity of illness, CGI-S,which is used to measure the severity of depressive, mania and severity overall. And, the UKU side-effects scale, which will assess all the side effects related or not to the study group treatments. In all visits, patients will be seen by the study psychiatrist and the research staff will complete mood ratings with the MADRAS, YMRS, CGI-BD, and the UKU side-effects scale.

At baseline (before randomization), week 8 and week 16 blood will be sampled for proinflammatory markers (C-reactive protein, soluble interleukin (IL)-2 receptor, IL-6 and tumor necrosis factor (TNF)-alpha), and oxidative stress markers (superoxide dismutase activity and catalase activity, serum thiobarbituric acid reactive substances (TBARS), which have been reported to be elevated in BD patients. These blood samples will be stored for possible future research on biomarkers or future genetic studies for up to 20 years, for use in pharmacogenetic research during this 20 year timeframe. The samples will be stored at the Wet Lab, in a double locked -80 degrees freezer, at BBSB, Department of Psychiatry at University of Texas Health Science Center at Houston. (1941 East Road, suite# 3170 Houston-TX 77054) for future use studying factors of Bipolar Disorder. When (or before) the 20 year period ends, the blood sample will be destroyed.

At the screening visit, week 8, and week 16 we will also be testing the Lithium levels in all patients that have been prescribed and currently taking the medication for study purposes. This extra test will be conducted for the safety of the patient and more Lithium level tests can be ordered under the PI's discretion throughout the 16 week trial.

Risks and potential benefits:

Aspirin is a safe medication for administration to humans and is approved by the FDA as an anti-inflammatory and analgesic agent. The dose proposed for this study is within the safety range as per medication package. Its side-effect profile is overall very favorable and it has met widespread use worldwide over the past decades. The main safety issues relate to the possibility of gastrointestinal complications, which are rare (and will be closely monitored in the weekly or biweekly visits that the study requires), and the propensity to interfere with coagulation and cause consequent bleeding (which will be prevented by excluding any individuals on use of anticoagulants or with active bleeding problems). There were a few case reports and small case series with other non-steroidal anti-inflammatory agents suggesting worsening of depressive symptoms related to treatment (e.g., indomethacin, ibuprofen, naproxen), but those were uncontrolled reports with individuals who suffered from other medical illnesses (rheumatologic diseases).

For our proposed trial, because some patients may be on lithium at the time they start on aspirin, we will exclude individuals with pre-existing cardiac and kidney disease. For patients on lithium, we will carefully monitor their serum lithium levels every two weeks during the course of the trial. Therefore, at the doses that are being proposed we do not anticipate any significant problems related to safety of the proposed intervention.

NAC is a safe compound that is commonly available and utilized over-the-counter. In a recent study the tolerability was excellent and main side effects included changes in energy level, headaches, heartburn and joint pain

Blood Draws: When the blood is drawn, there may be some minimal discomfort and/or bruising. Infection, excess bleeding, clotting, or fainting is also possible, although unlikely. All usual precautions will be taken to prevent these possibilities and these risks will be minimized by using trained staff to perform the blood draws

Subjects will be carefully monitored. If a subject's condition worsen to the point that he/she might become suicidal or severely depressed, we will terminate the subject's participation in the study and referred to his/her psychiatrist for psychiatric treatment.

Breach of Confidentiality: Every effort will be made to protect the subject identity and information during the study. All lab work and scan reports will be de-identified and the medical records will be protected. However, there is a small chance that the subject information may be viewed by someone that is not involved in the research study.

The study drug must be taken only by the person for whom it has been prescribed, and it must be kept out of the reach of children or persons of limited capacity to read or understand.

By sharing your sample with the study doctor, there is a risk of the possible loss of the subject privacy. Although no identifiable (name, address, etc.) information will be shared with others outside of this research project. The clinical information obtained from subjects will be part of their medical records and maintained at UT Center of Excellence on Mood Disorders, in the Department of Psychiatry at UTHSC-H, in facilities with adequate safeguards for the protection of confidentiality. The research data will be collected and recorded using only arbitrary code numbers for identification, in order to safeguard the confidentiality. All data will be kept in a secure area. Only the members of the UT Center of Excellence on Mood Disorders research group, who will get approval from CPHS, will have access to the data files, or to the master list for the codes. For publications purposes, the patients will be designated only by their assigned codes.

These blood samples, for use in pharmacogenetic research during this 15 year timeframe, samples will be stored at the Wet Lab, in a double locked -80 degrees freezer, at BBSB, Department of Psychiatry at University of Texas Health Science Center at Houston. (1941 East Road, suite# 3170 Houston-TX 77054) The possibility exists that the subject information may be taken and used for reasons outside of this project. The United States' Genetic Information Nondiscrimination, Act (GINA) of 2008, does not allow for employers or health insurance companies to discriminate against the research subject based on his/her genetic information. This means that health insurance companies or employers are NOT ALLOWED BY LAW to ask or use any of the subject genetic information (DNA, RNA, etc.) gained through testing to make decisions that affect the subject or hisher family's health coverage or income in a negative way

Importance of knowledge that may reasonably be expected to result:

The study will examine possible novel mechanism of actions with modulation of inflammatory mechanisms and oxidative stress and could result in the development of novel, low cost, safe and widely available treatments for BD patients who have not responded to other commonly utilized alternatives

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. A diagnosis of BD type I or II according to SCID-I interview;
3. Currently in a depressive or mixed episode, based on DSM-IV/ SCID-I criteria;
4. MADRAS >20 at entry in the study;
5. No CURRENT liver, kidney, heart disease or ulcers or bleeding dyscrasia;
6. No HYSTORY of kidney dysfunction or cardiac problems;
7. ON therapeutic doses of a mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations for at least ONE month.
8. Allowed psychiatric co-morbid conditions, such as anxiety disorders, PTSD and substance use (as long as do NOT meet abuse or dependence criteria according to the SCID-I in the past 2 months).

Exclusion Criteria:

1. CANNOT be on any :

   Anti-inflammatory: NSAIDs: Aspirin (bufferin, bayer aspirin, ecotrin), diflunisal (dolobid, diflunisal),Salsalate (amigesic, salflex), Ibuprofen (motrin, advil), Naproxen (naprosyn,aleve, midol extended relief), Fenoprofen (nalfon), Ketoprofen (actron), dexketoprofen(ketron D), Flurbiprofen (ansaid), Oxaprozin (daypro), Loxoprofen (loxfen, loxonin), Indomethacin (indocin, indocin SR), Sulindac (clinoril), Etodolac (lodine), Ketorolac (toradol), diclofenac (voltaren, cataflam), Nabumetone (Relafen) Piroxicam (feldene), Meloxicam (mobic), Tenoxicam (mobiflex), Lornoxicam (xefo),mefenamic acid (ponstel), meclofenamic acid (meclofenamate sodium), celecoxib (celebrex) Anticoagulants: Coumadin (Warfarin), Heparin Anti-oxidant agents Fish oil NAC ( N-acetyl cysteine)
2. Pregnancy
3. CANNOT change the dose of the psychotropic medications during the trial

Women Able to Become Pregnant: Participation in this study may involve risks to an embryo, fetus, or unborn child. If the subject is a female and able to become pregnant, a urine pregnancy test will be performed which must be negative prior to enrolling into the study, and the subject must agree not to become pregnant during the study. Urine pregnancy tests will be performed at Screening visit and week 8. The study staff will review adequate birth control methods with the subject and will remind her that she should not become pregnant during the study. Appropriate methods of birth control include: hormonal contraceptives (such as birth control pills, patches, and implants), barrier methods (such as a condom and diaphragms and spermicidal foam or jelly, surgical (hysterectomy or tubal ligation) or intrauterine device (IUD). The subject will be instructed to notify the study doctor immediately if there is a chance that she has become pregnant.

Also, if the subject is breast-feeding an infant or plan on breast-feeding an infant, she must notify the study doctor. It is not known if this drug is excreted in human milk; therefore, breast-feeding is not permitted during the study.

Patients can be on any mood stabilizing agents or combinations, as well as on other psychotropic medications at study entry, and the doses of those medications cannot be changed during the trial. They cannot be on any anti-inflammatory or anti-oxidant agents or anticoagulant at the point they are enrolled. If patients decompensate significantly, and/or become acutely suicidal, participation on the trial will be terminated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jair C Soares, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UT Center of Excellence on Mood Disorders, Houston, Texas, United States

REFERENCES:
- [Derived] Dean RL, Marquardt T, Hurducas C, Spyridi S, Barnes A, Smith R, Cowen PJ, McShane R, Hawton K, Malhi GS, Geddes J, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with bipolar disorder. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD011611. doi: 10.1002/14651858.CD011611.pub3. PMID 34623633
- [Derived] Bauer IE, Green C, Colpo GD, Teixeira AL, Selvaraj S, Durkin K, Zunta-Soares GB, Soares JC. A Double-Blind, Randomized, Placebo-Controlled Study of Aspirin and N-Acetylcysteine as Adjunctive Treatments for Bipolar Depression. J Clin Psychiatry. 2018 Dec 4;80(1):18m12200. doi: 10.4088/JCP.18m12200. PMID 30549489
- See also: UT Center of Excellence on Mood Disorders at Houston — https://med.uth.edu/psychiatry/research/centers/mood-disorders/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly assigned to one of the four arms during weeks 0-8. For patients who did not respond to treatment in period one, they were re-randomized to one of the other three arms and received a drug they had not yet received during period one. 8 were re-randomized to a different arm during period two.
Groups:
- Aspirin and NAC: research subject will be taking aspirin 1000mg (2 capsules of 500mg) every morning and NAC 1000mg (2 capsules of 500mg) two times a day in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations.
  Aspirin and NAC: aspirin 1000mg (2 capsules of 500mg) every morning and NAC 1000mg (2 capsules of 500mg) two times a day in addition to his/her antidepressant and/or mood stabilizer medicine
Period: Baseline Allocation
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Started | 5 | 9 | 9 | 15
Completed | 4 | 8 | 4 | 8
Not Completed | 1 | 1 | 5 | 7
Period: Week 8 Re-Randomization
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Started (Non-responders during Period 1 were re-randomized at week 8 into a new treatment arm.) | 4 (Non-responders during Period 1 were re-randomized at week 8 into a new treatment arm.) | 5 (Non-responders during Period 1 were re-randomized at week 8 into a new treatment arm.) | 5 (Non-responders during Period 1 were re-randomized at week 8 into a new treatment arm.) | 10 (Non-responders during Period 1 were re-randomized at week 8 into a new treatment arm.)
Completed | 4 | 5 | 4 | 7
Not Completed | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported using arm assignment for completers of period one. Patients were randomly assigned to one of four arms during period one, weeks 0-8. Patients who did not respond in period one were re-randomized during period two. Overall Number includes those withdrawn prior to week 8, so it is larger than the number analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill | Total
Number analyzed (Participants) | 4 | 8 | 4 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 4 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15.21) | 36.38 (7.05) | 40 (17.64) | 39.13 (9.99) | 40.56 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 6 | 15
  Male | 1 | 3 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 7 | 2 | 6 | 19
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 2 | 5 | 4 | 6 | 17
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 4 | 8 | 24
MADRS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10 item instrument with an overall score ranging from 0 to 54 points. A higher score corresponds with more severe depressive illness.
  units on a scale | 22.5 (10.47) | 19.38 (4.87) | 19.5 (1) | 22.88 (4.09) | 21.08 (5.45)
YMRS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) is an 11 item instrument with an overall score ranging from 0 to 60 points. A higher score corresponds with more severe manic illness.
  units on a scale | 4 (5.42) | 5.5 (3.46) | 5.75 (4.27) | 4.38 (4.63) | 4.92 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Demonstrating a > 50% Decrease in Depression Scores on the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The questionnaire includes questions on the following symptoms: 1. Apparent sadness; 2. Reported sadness; 3. Inner tension; 4. Reduced sleep; 5. Reduced appetite; 6. Concentration difficulties; 7. Lassitude; 8. Inability to feel; 9. Pessimistic thoughts; and 10. Suicidal thoughts.
Time Frame: Received drug for 8 weeks during week 0 to week 8 of the study
Measure: Count of Participants; unit: Participants
Groups:
- N-Acetyl Cysteine (NAC): Examine efficacy of NAC in treating depression in bipolar patients in a double-blind placebo-controlled add-on design. Proportion of patients demonstrating > 50% decrease in depression scores on the MADRS, as a Function of Treatment (on NAC treatment only). (We completed follow-up analyses with a 30% MADRS improvement criterion due to our limited sample size compared to original goals, as we fell short on patient recruitment goals and ended up with a somewhat underpowered study.)
- Placebo: research subject will be taking 4 capsules of matching sugar pill( placebo) in the morning and 2 capsules of matching placebo in the evenings in addition to his/her mood stabilizing drug (lithium, anticonvulsants, any atypical antipsychotics) or combinations
Arm/Group | Aspirin and NAC | Aspirin | N-Acetyl Cysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 4 | 8 | 8
Participants | 3 | 2 | 5 | 6

2. Primary Outcome: Number of Patients Demonstrating a > 50% Decrease in Depression Scores on the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 1
Time Frame: Received drug for 8 weeks during week 9 to week 16 of the study
Population: Patients who responded to treatment during week 0-8 were maintained on current treatment. Patients who did no respond were re-randomized for week 9-16.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin and NAC | Aspirin | N-Acetyl Cysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 4 | 5 | 7
Participants | 3 | 1 | 3 | 4

3. Primary Outcome: Number of Patients Demonstrating a > 30% Decrease in Depression Scores on the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The questionnaire includes questions on the following symptoms: 1. Apparent sadness; 2. Reported sadness; 3. Inner tension; 4. Reduced sleep; 5. Reduced appetite; 6. Concentration difficulties; 7. Lassitude; 8. Inability to feel; 9. Pessimistic thoughts; and 10. Suicidal thoughts. This 30% MADRS reduction was analyzed in addition to initial outcome measures of 50% MADRS reduction due to the smaller than expected study sample size.
Time Frame: Received drug for 8 weeks during week 0 to week 8 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin and NAC | Aspirin | N-Acetyl Cysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 4 | 8 | 8
Participants | 3 | 2 | 6 | 7

4. Primary Outcome: Number of Patients Demonstrating a > 30% Decrease in Depression Scores on the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 3
Time Frame: Received drug for 8 weeks during week 9 to week 16 of the study
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin and NAC | Aspirin | N-Acetyl Cysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 4 | 5 | 7
Participants | 4 | 3 | 3 | 4

5. Secondary Outcome: Inflammation as Indicated by C-reactive Protein (CRP) Levels
Description: C-reactive protein (CRP) levels are blood test markers of inflammation. Higher CRP corresponds with higher levels of inflammation. CRP is measured in milligrams per liter.
Time Frame: baseline, week 8, week 16
Population: Row numbers differ from overall number analyzed either due to patient withdrawal from study prior to completion, or from failure to obtain a blood sample from patient during study. Overall number analyzed differs from overall number of baseline participants for the same reason.
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 3 | 7 | 3 | 6
milligrams per liter
  CRP at Baseline | 6.85 (4.72) | 17.65 (13.51) | 5.1 (2.86) | 17.30 (20.74)
  CRP at Week 8: number analyzed (Participants) | 3 | 1 | 2 | 5
  CRP at Week 8 | 6.82 (8.4) | 41.09 (0) | 17.02 (9.21) | 7.4 (6.1)
  CRP at Week 16: number analyzed (Participants) | 3 | 6 | 2 | 6
  CRP at Week 16 | 10.76 (11.29) | 17.69 (10.98) | 9.39 (7.05) | 13.10 (17.98)

6. Secondary Outcome: Inflammation as Indicated by Interleukin 6 (IL-6) Levels
Description: Interleukin 6 (IL-6) is an interleukin that acts as a pro-inflammatory cytokine and an anti-inflammatory myokine. IL-6 is measured in picograms (pg) per milliliter (mL). Elevated interleukin-6 indicates potential immune system dysregulation and increased inflammation.
Time Frame: baseline, week 8, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 3 | 7 | 3 | 6
picograms per milliliter
  IL-6 at Baseline | 1.27 (.83) | 3.22 (2.02) | .85 (.79) | 2.3 (1.47)
  IL-6 at Week 8: number analyzed (Participants) | 3 | 1 | 2 | 5
  IL-6 at Week 8 | .78 (.43) | 3.53 (0) | 1.76 (.64) | 1.87 (.55)
  IL-6 at Week 16: number analyzed (Participants) | 3 | 6 | 2 | 6
  IL-6 at Week 16 | .90 (.57) | 2.6 (1.84) | 1.72 (1.15) | 1.71 (1.11)

7. Secondary Outcome: Inflammation as Indicated by Soluble Interleukin-2 (IL-2) Receptor Levels
Time Frame: baseline, week 8, week 16
Population: Data was not collected for this outcome measure. Blood samples were collected from participants, but tests for this particular outcome measure were not completed.
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Inflammation as Indicated by Tumor Necrosis Factor (TNF)-Alpha Levels
Time Frame: baseline, week 8, week 16
Population: as for outcome 7
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Oxidative Stress as Indicated by Superoxide Dismutase Activity
Time Frame: baseline, week 8, week 16
Population: as for outcome 7
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Oxidative Stress as Indicated by Catalase Activity
Time Frame: baseline, week 8, week 16
Population: as for outcome 7
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Oxidative Stress as Indicated by Serum Thiobarbituric Acid Reactive Substances (TBARS) Levels
Time Frame: baseline, week 8, week 16
Population: as for outcome 7
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during study participation - 16 weeks or until participants withdrew from the study.
Description: The number at risk for each arm includes the number at risk during week 0 to week 8 plus the number at risk during week 9 to week 16.
Arm/Group | Aspirin | N-acetyl-cysteine | Aspirin and NAC | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14 | 0/14 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14 | 1/14 | 1/25
Other Adverse Events (participants affected / at risk) | 1/9 | 0/14 | 1/14 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=9) | N-acetyl-cysteine (N=14) | Aspirin and NAC (N=14) | Sugar Pill (N=25)
Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Depression/Suicidal Ideations
Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Manic Episode of Bipolar I Disorder
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=9) | N-acetyl-cysteine (N=14) | Aspirin and NAC (N=14) | Sugar Pill (N=25)
Positive Pregnancy Test (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Positive pregnancy test at final study visit. All preceding pregnancy tests were negative throughout the study visits.
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Skin Irritation / Rash - Experience by a patient (determined likely due to citrus allergy) who was re-randomized after week 8. the same patient experienced the rash while taking Aspirin and then while on Placebo.

LIMITATIONS AND CAVEATS:
Mild to moderately severe depressive symptoms at baseline (therapeutic effects of NAC and Aspirin would have been different in more depressed sample). Small sample size (findings lack the required precision in estimates of effect).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT01797575/Prot_SAP_000.pdf